CLINICAL TRIAL: NCT06360952
Title: A Comparator Study of a Tasso Device to Traditional Venous Blood Sampling Methods for Complete Blood Count (CBC) With 5-part Differential in Patients With Leukemia, Lymphoma, and/or Other Blood Cell Disorders
Brief Title: A Comparator Study of a Tasso Device Blood Sample to Traditional Venous Blood Sample for CBC
Status: Not yet recruiting | Type: Observational
Sponsor: Tasso Inc. (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: T23-03
Record Dates: First submitted 2024-02-02; First posted 2024-04-11 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Leukopenia; Leukocytosis; Neutropenia
Keywords: leukocytosis; neutropenia; leukopenia; CBC; Tasso
MeSH Terms: conditions — Leukopenia; Leukocytosis; Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- leukopenia: Participants that have abnormal laboratory results for leukopenia. Participants will be assigned to all cohorts they have abnormal laboratory results for.
  Interventions: Device: Tasso+ CBC
- leukocytosis: Participants that have abnormal laboratory results for leukocytosis. Participants will be assigned to all cohorts they have abnormal laboratory results for.
  Interventions: Device: Tasso+ CBC
- neutropenia: Participants that have abnormal laboratory results for neutropenia. Participants will be assigned to all cohorts they have abnormal laboratory results for.
  Interventions: Device: Tasso+ CBC

INTERVENTIONS:
Device: Tasso+ CBC — Novel blood collection device

SUMMARY:
This study will evaluate the feasibility of using capillary blood samples collected with the Tasso device for analysis of CBC in diseased patients with leukemia, lymphoma, and/or other blood cell disorders.

This investigation will include a minimum of 40 sample sets from unique patients.

DETAILED DESCRIPTION:
This study will evaluate the feasibility of using capillary blood samples collected with the Tasso device for analysis of CBC in diseased patients with leukemia, lymphoma, and/or other blood cell disorders.

This investigation will include a minimum of 40 sample sets from unique patients.

The primary aim of this study is to demonstrate the agreement between capillary blood collected using the Tasso device and venous blood collected in a K2EDTA (dipotassium ethylenediaminetetraacetic acid) tube according to established sampling procedures for quantification of WBC and ANC as part of a standard CBC panel with 5-part differential.

The secondary aim of the study is to demonstrate the agreement between Tasso device and venous samples for the measurement of additional analytes evaluated as part of a standard CBC panel with 5-part differential, including PLTs, HGB, RBC, Hct, MCV, lymphocytes, monocytes, eosinophils, and basophils.

An exploratory aim of this research is to evaluate patient acceptance of the Tasso device in a diseased population.

Adverse Events (AEs) occurring up to 24 hours after use of the Tasso device will be evaluated.

Patient response to using the Tasso device will be collected via simple survey.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written (or electronic) informed consent prior to study entry
2. At least 18 years of age
3. Requiring a CBC blood test as part of the patient's standard of care
4. Have abnormal laboratory results of either leukopenia, leukocytosis or neutropenia.
5. Normal skin integrity and healthy skin appearance around the capillary collection site (upper arm/shoulder area on at least one side)

Exclusion Criteria:

1. Unable to give full and free consent to participate in a study due to limited capacity or risk of undue influence or coercion (including but not limited to children, prisoners, individuals with diminished decision-making capacity, illiterate or educationally disadvantaged populations) or any other individual who is unable to give full and free consent in the judgement of the investigator
2. At the determination of the treating physician, unsuitable for enrollment due to severe immunocompromised status or other comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known blood cancers and/or blood cell disorders resulting in abnormal laboratory results for either leukopenia, leukocytosis or neutropenia will be recruited and enrolled into this study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between capillary and venous blood in the measurement of White Blood Cells and Absolute Neutrophil Count | Day 1
  To demonstrate agreement between capillary blood collected using the Tasso device and traditional venous blood collected using standard methods for measurement of white blood cells (WBCs), and absolute neutrophils count (ANC) as part of a CBC analysis with 5-part differential.

SECONDARY OUTCOMES:
Agreement between capillary and venous blood in the measurement of secondary biomarkers | Day 1
  To demonstrate agreement between capillary blood collected using the Tasso device and traditional venous blood collected using standard methods for measurement of remaining CBC components including platelets (PLTs), hemoglobin (HGB), red blood cells (RBCs), hematocrit (Hct), and mean corpuscular volume (MCV), as well as differential quantification of lymphocytes, monocytes, eosinophils, and basophils.

OTHER OUTCOMES:
Patient acceptance of Tasso device | Day 1
  To evaluate patient acceptance of the Tasso device in a diseased population via survey responses. Survey responses will consist of a series of questions referencing the participant perception of the experience with the Tasso device using The Satisfaction Scale under the parameters of 1 through 5 (1 - Strongly Disagree through 5 - Strongly Agree) and other questions asking for participant preference in regards to the means of sample collection and location (ex. Venipuncture versus Tasso, self-collected at home or preformed at a doctor's office or clinic).

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Berthier, Phd, Principal Investigator — Tasso Inc.
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No